CLINICAL TRIAL: NCT05219279
Title: Novel Radial Diffusion-Weighted MR Spectroscopic Imaging of HIV: Biomarker Detection Using Functional Imaging and Neurocognitive Correlates
Brief Title: MR Imaging and MR Spectroscopy of HIV
Acronym: HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Michael Albert Thomas, Ph.D., Professor-in-Residence, University of California, Los Angeles
Other Study IDs: 20-001739
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
Keywords: MR Spectroscopy; central nervous system
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV+ participants: * HIV-infected between age of 20 and 65 years
  * Consistently have plasma HIV RNA levels <200 copies/mL for at least the last 12 months on a stable antiretroviral regimen with any changes made only for convenience, safety or simplicity.
- HIV- participants: 25 age- and sex- matched HIV- subjects (healthy) will be recruited also at the UCLA Medical center who will undergo the neuroimaging examination.

SUMMARY:
The Center for Disease Control and Prevention estimates that 1,148,200 Americans aged 13 years and older are living with HIV infection, including 207,600 (18.1%) who are unaware of their infection. According to pathological data, central nervous system (CNS) involvement is commonly found during the early phase of infection. In vivo proton magnetic resonance spectroscopy studies of HIV-infected humans have demonstrated significant changes of metabolites observed in the brain N-acetylaspartate, creatine, choline, glutamate, glutamine and myo-inositol with varying changes in different brain regions. Diffusion tensor imaging (DTI) is a novel functional MRI technique which can be used to derive quantitative in vivo measurements of region-specific and diffuse brain alterations. DTI studies have demonstrated changes of mean diffusivity (MD) and fractional anisotropy (FA) in the various parts of brain. Diffusion abnormalities involving various regions of brain have also been observed in patients infected with HIV. One dimensional (1D) or two-dimensional (2D) magnetic resonance spectroscopic imaging (MRSI) technique has been used for many years to study the metabolites changes in HIV. MRI scan time necessary for the acquisition of high-resolution MRSI data with adequate spatial coverage may be prohibitively long for clinical exams. Thus, new imaging and bio-chemical characterization techniques are needed to allow repeated, non-invasive assessment of these processes in vivo. Since neuroinflammation is associated with increased brain water, diffusion tensor imaging (DTI) is sensitive to changes in white matter (WM) and inflammatory changes associated with HIV infections. Even though only single-voxel-based diffusion-weighted MRS has been previously investigated, altered diffusivity of non-water metabolites and its relationship with metabolic disturbance as well as structural and functional abnormalities in HIV has not been investigated. The brain apparent diffusion coefficient (ADC) changes of metabolites measured by the novel 3D MRSI technique will be correlated with the ADCs and fractional anisotrophy of water recorded by DTI and cell count to better understand the role of CNS involvement in HIV pathology.

DETAILED DESCRIPTION:
This will be a multicenter prospective study. We will recruit ten (10) healthy participants aged 20 to 30 years to investigate the feasibility and test/retest reliability of the REPSI sequence. Twenty five (25) HIV+ patients will be recruited from the Division of HIV Medicine (Dr. Eric Daar) at the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center (Torrance, CA). HIV+ patients will be transported to the UCLA Medical center for neuroimaging examination.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected between age of 20 and 65 years
* Consistently have plasma HIV RNA levels <200 copies/mL for at least the last 12 months on a stable antiretroviral regimen with any changes made only for convenience, safety or simplicity.
* Able to provide informed consent.

Exclusion Criteria:

-HIV negative

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 HIV-infected, virologically suppressed and 25 age- and sex- matched HIV- subjects (healthy) will be recruited also at the UCLA Medical center who will undergo the neuroimaging examination.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-07-09 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Spectroscopy outcomes | One year
  (1) Develop accelerated r-DW-EPSI using semi-LASER localization (33), and optimize the protocol in brain phantom solutions and 10 healthy adults. (2) Determine ADCs of Cr, NAA, Cho, mI and Glx in 25 adult HIV patients on ART, and evaluate differences in 25 age-/sex-matched HIV- adults. Outcomes will be correlated with DTI metrics, neuropsychological test results, and other disease variables

CONTACTS AND LOCATIONS:
Overall Officials: Albert Thomas, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States